CLINICAL TRIAL: NCT00501995
Title: High Dose Cyclophosphamide for Treatment of Systemic Sclerosis (Scleroderma)
Brief Title: High Dose Cyclophosphamide for Treatment of Scleroderma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Fredrick M. Wigley, Professor of Medicine, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-11-17-02
Record Dates: First submitted 2007-07-13; First posted 2007-07-17 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Scleroderma
Keywords: High Dose Cyclophosphamide; Systemic Sclerosis; Scleroderma; immunoablation
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IV Cyclophosphamide (50 mg/kg) (Experimental): This is an open-labeled single arm study of Cyclophosphamide (50 mg/kg) administered intravenously over 1 hour daily for four consecutive days (200 mg/kg total) through a Hickman catheter .
  Interventions: Drug: IV Cyclophosphamide

INTERVENTIONS:
Drug: IV Cyclophosphamide — Cyclophosphamide (50 mg/kg) intravenously daily for 4 consecutive days (total 200 mg/kg) followed by granulocyte colony-stimulating factor (5 µg/kg/day)
  Other Names: Cytoxan, Neosar

SUMMARY:
Systemic Sclerosis (Scleroderma) varies greatly in clinical manifestations, mode of presentation, and course. The natural history of this chronic autoimmune disease ranges from benign to fatal. Patients are classified into limited and diffuse scleroderma defined by the degree of skin involvement. Patients with limited disease (e.g. the C.R.E.S.T. syndrome) generally have mild disease and normal survival. However, patients with diffuse cutaneous scleroderma often have severe multi-system disease that is not only devastating emotionally and physically but is associated with a 60-70% five year survival and a 40-50% 10 year survival. No therapies have proven effective in the treatment of scleroderma. Strategy to treat scleroderma have included attempts to prevent fibrosis with drugs that interfere with collagen metabolism, attempts to modify the disease process by immunosuppression and attempts to alter the disease by vasoactive drugs. High dose of corticosteroids and other immunosuppressive drugs (e.g. chlorambucil, 5-fluorouracil, methotrexate, cyclophosphamide, cyclosporine) used at conventional doses have not proven curative, but have shown some benefit for inflammatory features of the disease (e.g. arthritis, myositis, fibrosing alveolitis).

Both allogeneic and autologous bone marrow transplantation (BMT) have shown to modify and in some instances reverse a variety of animal models of autoimmune disease. This has prompted many investigators to propose the use of peripheral blood stem cell transplantation (PBSCT) for the treatment of autoimmune disease including scleroderma. Unfortunately, this approach risks infusing untreated autoreactive lymphocyte clones after the immunoablative preparative regimen. We have previously demonstrated that high-dose cyclophosphamide without BMT can induce durable and complete remissions in another autoimmune disease, severe aplastic anemia. Recent data with high dose cyclophosphamide show that it can induce complete remissions in other autoimmune hematologic disorders. The objective of this study is to determine whether high dose cyclophosphamide can induce a durable remission in scleroderma patients with life-threatening disease, and to determine toxicity of high dose cyclophosphamide in high risk scleroderma patients.

DETAILED DESCRIPTION:
Study design

The study was an open-label, single-site trial of a single exposure to high-dose cyclophosphamide without stem cell rescue. Each patient was followed up by the same doctor to eliminate interobserver skin score variation. Baseline measurements included comprehensive laboratory studies that included complete blood count with differential, comprehensive metabolic panel, urine analysis with culture, quantitative immunoglobulins, antibodies to hepatitis B core and surface antigens and antibodies to hepatitis C, human immunodeficiency, herpes, varicella, Epstein-Barr viruses; rapid plasma reagin test, chest x-ray or high-resolution computed tomography (HRCT) scan of the lungs, pulmonary function testing, electrocardiogram, and echo or multigated acquisition (MUGA) scan.

The primary clinical efficacy end point was the modified Rodnan skin score (mRSS).24 A 25% sustained improvement in the mRSS at any point in the follow-up was considered clinically important and a successful outcome.25 Secondary outcome measures included the Health Assessment Questionnaire-Disability Index (HAQ-DI) and physician global assessment (PGA) determined by a visual analogue scale on a scale from 0 to 100. Values for the percentage predicted lung volumes were referenced from NHANES/Hanikson et al26 and for diffusing capacity of the lungs for carbon monoxide (DLCO) from Knudson et al.27 The disease duration was defined as the time from the first non-Raynaud's symptom related to scleroderma to study entry.

Treatment protocol

Cyclophosphamide (50 mg/kg) was administered intravenously over 1 hour daily for four consecutive days (200 mg/kg total) through a Hickman catheter. The dose of cyclophosphamide was based on the ideal body weight as determined by the Metropolitan Life tables.28 29 If the patient's actual weight was less than the ideal body weight, the actual body weight was used to calculate the cyclophosphamide dose. Intravenous mesna (10 mg/kg) was given 30 minutes before cyclophosphamide and then 3, 6 and 8 hours after cyclophosphamide was administered for prophylaxis against haemorrhagic cystitis. Intravenous ondansetron (32 mg) was administered 1 hour before each dose of cyclophosphamide. Six days after the last dose of cyclophosphamide, all patients received granulocyte colony-stimulating factor (5 µg/kg/day) until the neutrophil count was 1×109/l for two consecutive days. Prophylactic antibiotic support, consisting of fluconazole (400 mg/day), norfloxacin (400 mg/day), and valaciclovir (500 mg twice a day, if antibodies to herpes simplex were present), was given beginning the day after the last dose of cyclophosphamide and continuing until the neutrophil count exceeded 0.5×109/l. Dapsone (100 mg three times a week for 6 months) or trimethoprim-sulfamethoxazole (80/400 mg three times a week for 6 months) was administered for Pneumocystis carinii prophylaxis. Packed red blood cell (leucocyte-poor) transfusions were administered to maintain a haematocrit level >25%. Platelet transfusions were given for bleeding or to maintain a platelet count >10×109/l, or both. All blood products were irradiated (>2000 rad) to prevent graft versus host disease.

ELIGIBILITY:
Inclusion Criteria:

* Meet established criteria for a diagnosis of diffuse cutaneous scleroderma and have evidence of moderately severe organ damage and clinical evidence of active disease.
* Patients with diffuse scleroderma who have evidence of active fibrosing alveolitis manifested by either a greater than 10% decline in the forced vital capacity or the diffusing capacity from the defined normal values or from baseline measurements.
* Patients with severe deforming localized scleroderma (generalized morphea, liner morphea, keloid or bullous scleroderma) that threatens their capacity to function normally in society.

Exclusion Criteria:

* Age less than 18 years and over 70 years
* Any risk of pregnancy
* Cardiac ejection fraction of < 45%
* Serum creatinine > 3.0
* Patients who are pre-terminal or moribund
* Bilirubin > 2.0, transaminases > 2x normal
* Forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), (5/30/01) < 50% predicted

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2001-02; Primary Completion 2008-07 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fredrick M Wigley, MD, Principal Investigator — Johns Hopkins University

REFERENCES:
- [Result] Tehlirian CV, Hummers LK, White B, Brodsky RA, Wigley FM. High-dose cyclophosphamide without stem cell rescue in scleroderma. Ann Rheum Dis. 2008 Jun;67(6):775-81. doi: 10.1136/ard.2007.077446. Epub 2007 Nov 1. PMID 17974598

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV Cyclophosphamide (50 mg/kg)
Started | 6
Completed | 5
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Patients with scleroderma were considered eligible for this open-label trial if they had a diagnosis of diffuse cutaneous scleroderma and evidence of clinically active disease.
Groups:
- IV Cyclophosphamide (50 mg/kg): This is an open-labeled single arm study of Cyclophosphamide (50 mg/kg) administered intravenously IV Cyclophosphamide: Cyclophosphamide (50 mg/kg) intravenously daily for 4 consecutive days (total 200 mg/kg) followed by granulocyte colony-stimulating factor (5 µg/kg/day)
Arm/Group | IV Cyclophosphamide (50 mg/kg)
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 39 [19 to 60]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants] — Number of participants
  participants
    United States | 6
Number of Participants with diagnosis of scleroderma [Number; unit: participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Improvement in the Modified Rodnan Skin Score.
Description: The modified Rodnan skin score is the accepted clinical measure of scleroderma skin activity. The investigator will assess the thickening of the skin using the modified Rodnan skin score through simple palpation on 17 different body areas: fingers, hands, forearms, arms, feet, legs, and thighs (bilaterally) and face, chest, and abdomen (singly). Skin thickness is assessed on a scale of 0-3; 0 representing normal skin and 3 being severe thickening. The sum of the individual scores can range from 0-51; 0 (normal) to 51 (severe thickening in all 17 areas) A 25% improvement in the modified Rodnan Skin score will be considered significant at any time point in the study. Modified Rodnan Skin Score was evaluated at months 0,1,3,6,12 and 24 months.
Time Frame: 0 to 24 months
Population: Patient 4 died during the early phase of the study and longitudinal assessment of his skin score was not determined.
Measure: Mean (Full Range); unit: percent improvement from baseline
Arm/Group | IV Cyclophosphamide (50 mg/kg)
Number analyzed (Participants) | 5
percent improvement from baseline | 46.75 [31 to 60]

2. Secondary Outcome: Change in the HAQ-DI, PGA, FVC and DLCO
Description: The Health Assessment Questionnaire-Disability Index (HAQ-DI) a 48 item questionnaire assessing ability to perform activities of daily living, use of assistive devises and a 6 item analog scale of pain severity from 0 cm (no pain) to 14.3 cm (very severe pain). The lower the HAQ-DI score the less the disability. The physician global assessment (PGA) which is a visual analogue scale from 0 to 100 on which the physician rates the patient's disease severity based on their observations. A score of 0 is no disease activity and 100 is the worst possible disease activity. The Forced Vital Capacity (FVC) measure of lung capacity and Diffusing Capacity (DLCO) measures of oxygen exchange in the alveoli ( pulmonary function testing). The predicted lung volumes were referenced from NHANES/Hanikson et al and for DLCO predicts were from Knudson. Pre and post study percent predicted values were compared.
Time Frame: 0-24 months
Population: The study group consisted of 4 men and 2 women aged 19-60 years of old.
Measure: Mean (Full Range); unit: percentage change
Arm/Group | IV Cyclophosphamide (50 mg/kg)
Number analyzed (Participants) | 6
percentage change
  HAQ-DI score | 79 [0 to 93]
  PGA | 71 [62 to 80]
  FVC | 0 [-7 to 5]
  DLCO | 14 [2 to 29]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | IV Cyclophosphamide (50 mg/kg)
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Cyclophosphamide (50 mg/kg) (N=6)
Death (Infections and infestations) | 1 (1) — An infection leading to death within 8 weeks after cyclophosphamide therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Cyclophosphamide (50 mg/kg) (N=6)
neutropenic fever (Immune system disorders) | 5 (5)
nausea/vomitting (Gastrointestinal disorders) | 3 (3)
diarrhea (Gastrointestinal disorders) | 3 (3)
oedema (Vascular disorders) | 3 (3)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
septic bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 2 (2)
sexual dysfunction (Reproductive system and breast disorders) | 3 (3)
amenorrhea (Reproductive system and breast disorders) | 1 (1)
itch (Skin and subcutaneous tissue disorders) | 2 (2)
myalgias (Musculoskeletal and connective tissue disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
blurred vision (Eye disorders) | 1 (1)
alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
anaemia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No